CLINICAL TRIAL: NCT00884663
Title: Candesartan vs Propranolol for Migraine Prevention: A Double Blind, Placebo Controlled, Double Dummy, Triple Cross-over Study
Brief Title: Candesartan Versus Propranolol for Migraine Prevention
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: AstraZeneca (Industry); St. Olavs Hospital (Other); Kragerø Tablettproduksjon as, Norway (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-47-7006-2008; 2008-002312-17 (EudraCT Number)
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Migraine Without Aura; Migraine With Aura; Chronic Migraine
MeSH Terms: conditions — Migraine without Aura; Migraine with Aura | interventions — candesartan; Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Candesartan (Experimental)
  Interventions: Drug: Candesartan
- 2 propranolol (Active Comparator)
  Interventions: Drug: propranolol
- 3 Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Candesartan — Candesartan cilexitil tablets, 16 mg once daily
  Arms: 1 Candesartan
Drug: propranolol — Propranolol hydrochloride capsules 160 mg once daily, slow release formulation
  Arms: 2 propranolol
Drug: placebo — placebo tablets and capsules
  Arms: 3 Placebo

SUMMARY:
The main aim of the present study is to compare candesartan with propranolol for migraine prophylaxis.

DETAILED DESCRIPTION:
Candesartan was shown to be effective for migraine prophylaxis in a randomized double blind cross-over study published in 2003. The drug is now widely used for this purpose in many countries, although no confirmatory study has been published. The aims of the present study are: 1) to see if the results in the first candesartan study can be replicated in a new patient population, including patients with chronic migraine, and, 2) to perform a head-to-head comparison of candesartan 16 mg/day with standard treatment with propranolol 160 mg slow release. We also intend to study whether responsiveness to these drugs may be related to heart rate variability and baroreceptor sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* retrospectively have ≥ 2 migraine attacks per month during the last 3 months
* during the baseline period have ≥ 2 migraine attacks
* debut of migraine at least one year prior to inclusion
* start of migraine before age 50 years.

Exclusion Criteria:

* interval headache not distinguishable from migraine
* chronic tension-type headache or other headache occurring on ≥ 15 days/month
* pregnancy, nursing or inability to use contraceptives
* heart conduction block on ECG or significant ECG abnormality on inclusion
* heart rate < 54 after 3 minutes rest
* previous or present asthma, diabetes; decreased hepatic or renal function
* hypersensitivity to active substance
* history of angioneurotic edema
* significant psychiatric illness
* use of daily migraine prophylactics less than 4 weeks prior to start of study
* having tried ≥ 3 prophylactic drugs against migraine during the last 10 years
* previous use of propranolol or candesartan in adequate doses
* previous discontinuation of either Atacand or Inderal Retard (or another beta blocker) due to side effects
* current use of antihypertensive medication
* require use of rizatriptan (Maxalt) 10 mg tabl.
* subjects requiring detoxification from acute medication (ergotamines, opioids)
* patients who consistently fail to respond to any acute migraine medication
* patients with alcohol or illicit drug dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The number of days per 4 weeks with moderate or severe headache lasting ≥ 4 hours or is treated with the patient's usual headache medication | One year

SECONDARY OUTCOMES:
Days with headache | One year
Hours with headache | One year
Headache intensity (0-3 scale) on days with headache | one year
Doses of analgesics | one year
Doses of triptans | One year
Days with sick leave | one year
Number of responders (≥ 50% decrease in migraine days compared with baseline) | one year
Number of reported side effects | one year
Number of predefined retrospective side effects | one year

CONTACTS AND LOCATIONS:
Overall Officials: Lars J Stovner, Ph.D., Principal Investigator — Norwegian National Headache Centre, St. Olavs Hospital; Lars J Stovner, Ph.D., Study Director — Norwegian National Headache Centre
Locations (1):
- Norwegian National Headache Centre, St. Olavs University Hospital, Trondheim, Norway

REFERENCES:
- [Background] Tronvik E, Stovner LJ, Helde G, Sand T, Bovim G. Prophylactic treatment of migraine with an angiotensin II receptor blocker: a randomized controlled trial. JAMA. 2003 Jan 1;289(1):65-9. doi: 10.1001/jama.289.1.65. PMID 12503978
- [Result] Stovner LJ, Linde M, Gravdahl GB, Tronvik E, Aamodt AH, Sand T, Hagen K. A comparative study of candesartan versus propranolol for migraine prophylaxis: A randomised, triple-blind, placebo-controlled, double cross-over study. Cephalalgia. 2014 Jun;34(7):523-32. doi: 10.1177/0333102413515348. Epub 2013 Dec 11. PMID 24335848